CLINICAL TRIAL: NCT06147401
Title: Pericapsular Nerve Group (PENG) Associated with Lateral Femoral Cutaneous Nerve (LFCN) Block Versus FIC Block for Total Hip Replacement Surgery: a Double Blind Randomized Controlled Trial
Brief Title: Comparison of PENG Associated with LFCN Block Versus FICB for Multimodal Analgesic Management in THA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale Edoardo Bassini (Other)
Responsible Party: Principal Investigator, Francesco Vetrone, MD, Principal Investigator, Ospedale Edoardo Bassini
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3703
Record Dates: First submitted 2023-11-17; First posted 2023-11-27 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Regional Anesthesia Morbidity; Arthropathy of Hip; Hip Arthropathy; Post Operative Pain; Anesthesia Complication
Keywords: ERAS; Postoperative muscle weakness; Regional Block; Post Operative Analgesia
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: A double-blind, randomized, controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The anesthetist in the operating room will be the only one who knows what treatment has been administered
  Participant: the patient will not know the type of block he will be subjected to, because of he will already be subjected to neuraxial anesthesia.
  Outcomes Assessor: a clinician external to the practice will evaluate the degree of residual paralysis after anesthesia and pain control Investigator: the statistician will not know which anesthetic technique was administered to which group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PENG - LFCN Block (Experimental): group in which PENG and LFCN Block was performed. After performing neuraxial anesthesia, the PENG associated with LFCN block will be performed. Under ultrasound guidance, 20ml and 5ml of Ropivacaine 0.5% will be administered respectively.
  Interventions: Procedure: PENG plus LFCN block
- FIC Block (Active Comparator): group in which FIC Block was performed After performing neuraxial anesthesia, FIC block will be performed. Under ultrasound guidance, 20 ml of Ropivacaine 0.5% will be administered.
  Interventions: Procedure: FIC Block

INTERVENTIONS:
Procedure: PENG plus LFCN block — The experimental arm will be subjected to a combination of peripheral blocks: the interfascial block of the PENG and the perinervous block of the LFCN
  The PENG block involves deposition of local anesthetic in the fascial plane between the psoas muscle and the superior pubic ramus.
  The LFCN block consists of applying local anesthetic near the nerve. The LFCN lies in the subcutaneous plane deep to the fascia lata below the anterior superior ischiatic spine.
  Other Names: Pericapsular nerve group block and lateral femoral cutaneous nerve block; PENG and lateral femoral cutaneous nerve block
  Arms: PENG - LFCN Block
Procedure: FIC Block — The control arm will be subjected to an interfascial block, the fascia iliaca Compartment Block.
  The FICB consists in the injection of anaesthetic agents into the fascia iliaca compartment.
  Other Names: Fascia Iliaca Compartment Block; FICB
  Arms: FIC Block

SUMMARY:
Optimal pain control with limited muscle weakness is paramount for a swift initiation of physical therapy and ambulation. Fascia iliaca compartment block (FIC) has been recommended since it offers the best pain control with low risk of motor block. Pericapsular nerve group block (PENG) with lateral femoral cutaneous block (LFCN) has been proposed as an effective alternative to FIB that offers similar pain control with a considerably lower risk of motor block. The aim of this study is to compare the afore mentioned blocks and determine which one yielded the least degree of quadriceps femoris muscle weakness and the better pain control (the lowest NRS score with least need for opioids).

DETAILED DESCRIPTION:
This single-center, double blinded RCT investigation will be conducted at ASST Nord Milano - Bassini hospital. The study was approved by the ethics committee "Comitato Etico Territoriale Lombardia 3".

Each patient undergoing elective total hip replacement surgery with anterior approach will be subjected (unless contraindicated) to subarachnoid neuraxial anesthesia and immediately afterwards to a peripheral analgesic block: the FIC block or the association of PENG and FCLN block. The choice of block type will be randomized.

At the end of the procedure, a clinician unaware of the anesthetic technique used will assess the degree of residual motor block. Simultaneously, he will assess pain control in terms of NRS (Numerical Rating Scale) and the need for opioid use.

ELIGIBILITY:
Inclusion Criteria:

* elective total hip replacement surgery for non-traumatic hip disease,
* THA (total hip arthroplasty) with lateral approach
* age >18 years,
* signed consent form for spinal anesthesia and peripheral nerve block provided by the patient or legal guardian if appointed

Exclusion Criteria:

* Non elective THA
* Lack of consent to the procedure
* Contraindications to performing neuraxial anesthesia (i.e. Signs suggestive of puncture site infection, INR > 1.5, aPTT > 1.5, PLT < 40.000)
* Documented or suspected allergy to local anesthetics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
MRC at 6h | six hours after performing the regional anesthesia technique
  evaluation of the degree of weakness or residual paresis of the quadriceps femoris muscle on the operative side using 'the Oxford Scale' (aka Medical Research Council Manual Muscle Testing scale or MRC scale) The MRC scale is a 0-5 scale, with zero meaning "no contraction " and five meaning "Full range of motion against gravity with full resistance".
MRC at 24h | 24 hours after performing the regional anesthesia technique
  evaluation of the degree of weakness or residual paresis of the quadriceps femoris muscle on the operative side using 'the Oxford Scale' (aka Medical Research Council Manual Muscle Testing scale or MRC scale) The MRC scale is a 0-5 scale, with zero meaning "no contraction " and five meaning "Full range of motion against gravity with full resistance".
MRC at 48h | 48 hours after performing the regional anesthesia technique
  evaluation of the degree of weakness or residual paresis of the quadriceps femoris muscle on the operative side using 'the Oxford Scale' (aka Medical Research Council Manual Muscle Testing scale or MRC scale) The MRC scale is a 0-5 scale, with zero meaning "no contraction " and five meaning "Full range of motion against gravity with full resistance".

SECONDARY OUTCOMES:
time to first postoperative ambulation | From date of surgery until up to 72 hours after
  we studied the effect or Regional anesthesia on residual paralysis
Pain control at 6h | six hours after performing the regional anesthesia technique
  pain assessment with Numeric Rating Scale (NRS): a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable"
Pain control at 24h | 24 hours after performing the regional anesthesia technique
  pain assessment with Numeric Rating Scale (NRS): a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable"
Pain control at 48h | 48 hours after performing the regional anesthesia technique
  pain assessment with Numeric Rating Scale (NRS): a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable"
MME of PRN opioid total doses | From date of surgery until up to 72 hours after
  Morphine Milligram Equivalents (MME) of "pro re nata" (PRN) opioid total doses we will study the effect of Regional anesthesia on opioid-sparing with the same pre-established pain relief protocol
time to first PRN opioid request | From date of surgery until up to 72 hours after
  time to first PRN (pro re nata) opioid request expressed in minutes
need for PRN opioid | From date of surgery until up to 72 hours after
  number of opioid administration

OTHER OUTCOMES:
Complication | From date of surgery until up to 72 hours after
  any complications recorded in the first 72 hours including but not limited to: postoperative nausea and vomiting (PONV), vascular puncture, paresthesia and LA toxicity
the degree of hip flexion | six hours after performing the regional anesthesia technique
  Hip flexion degree of the operative side is measured using Digital Angle Gauge in supine position
the degree of hip flexion | 24 hours after performing the regional anesthesia technique
  Hip flexion degree of the operative side is measured using Digital Angle Gauge in supine position
the degree of hip flexion | 48 hours after performing the regional anesthesia technique
  Hip flexion degree of the operative side is measured using Digital Angle Gauge in supine position

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Edoardo Bassini, Cinisello Balsamo, Milano, Italy

IPD SHARING:
Plan to Share IPD: Undecided